CLINICAL TRIAL: NCT05156957
Title: Effect of Physiotherapy in Patients Presenting to the Emergency Department With Nonspecific Lower Back Pain. A Brief Intervention Focusing on Patient Reported Outcomes
Brief Title: Effect of Physiotherapy in Patients Presenting to the Emergency Department With Nonspecific Lower Back Pain
Acronym: EPAC-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-02166; am21Bingisser
Record Dates: First submitted 2021-11-29; First posted 2021-12-14 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Lower Back Pain
Keywords: physiotherapy intervention; Oswestry Disability Index (ODI); nonspecific lower back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The study intervention is a brief physiotherapeutic assessment, a brief information on the expected course of the condition, and a brief instruction on self-management, including three exercises for daily self-guided therapy.
  Interventions: Other: physiotherapeutic intervention
- control group (No Intervention): The control group will receive written information on the expected course of the condition, written instructions on self-management and written instructions on exercises for daily self-guided therapy.

INTERVENTIONS:
Other: physiotherapeutic intervention — The intervention consists of a brief physiotherapeutic assessment by a short physical performance battery, a brief information on the expected course of the condition and instructions on self-management regarding back friendly behaviour (eg. respecting the pain, staying active and back friendly movement strategies). Additionally, three exercises for daily self-guided therapy are included to the intervention: Turning in bed and coming to a sitting position, sit to stand and squats standing in front of a wall.
  Arms: intervention group

SUMMARY:
Physiotherapy is a long established therapy in lower back pain. It is unknown if physiotherapeutic interventions in patients presenting to the Emergency Department (ED) with nonspecific lower back pain are beneficial. The aim of this study is to assess whether patients presenting to the emergency department with non-specific low risk low back pain would benefit from a physiotherapy intervention, as compared to patients without physiotherapy intervention at time of ED presentation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Experiencing nonspecific lower back pain
* Presentation to the Emergency Department (ED) of the University Hospital Basel

Exclusion Criteria:

* Inpatient disposition after ED work-up
* "Red Flags" at time of ED-presentation:

  1. Major trauma in all patients
  2. Fractures leading to immobilization
  3. Severe or progressive sensory alteration or weakness
  4. Bladder or bowel dysfunction
  5. Evidence of neurological deficit on physical examination
  6. Severe chronic disease, such as metastasized cancer, palliative care
* Epidural steroid injections in the last 3 months
* Inability or contraindications to undergo the investigated intervention or to follow the study procedures, e.g. due to certain neurological disorders, language problems, psychological disorders, cognitive impairment, physical inability etc.
* Prior enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | At Day 0 and at Day 7 ± 7 days
  This self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Pain Numeric Rating Scale (NRS) | At Day 0, Day 7 ± 7 days, Day 21 ± 3 days, Day 42 ± 3 days
  The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain ('0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine"))
Feasibility of the intervention | At Day 0
  The questionnaire was completed by the physiotherapist after the intervention and consisted of six questions about the feasibility of the physiotherapeutic intervention. Each question had a scale of 1 (= no, strongly disagree) to 6 (=yes, strongly agree) for possible answers.
Patient satisfaction | At Day 7 ± 7 days
  This self-completed questionnaire contains six questions about patient satisfaction with their ED visit on day 0. Each question could be answered with a score from 0 (not at all) to 10 (very much).
Adherence to therapy recommendations | At Day 7 ± 7 days
  Patients were asked if they were able to adhere to the behavioral and exercise recommendations given to them on Day 0.
StarT Back Screening Tool (SBST) | Day 0, Day 7 ± 7 days, Day 42 ± 3 days
  The SBST categorises back pain patients into 3 categories: low, medium and high risk. It consists of 9 items, each with a value of 0 or 1 points. The SBST Score is calculated by summing the points from each question, with a minimum score of 0 points and a maximum score of 9 points.
Oswestry Disability Index (ODI) | Day 21 ± 3 days, Day 42 ± 3 days
  This self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Pain medication use | At Day 0, Day 7 ± 7 days, Day 21 ± 3 days, Day 42 ± 3 days
  Questions about the use of pain medication and how long pain medication have been used.
Utilization of medical resources | At Day 7 ± 7 days, Day 21 ± 3 days, Day 42 ± 3 days
  Patients were asked if they had seen a physiotherapist, an emergency department, a general practitioner, a specialist, been hospitalized or had imaging since the last contact.
Ability to work | At Day 7 ± 7 days, Day 21 ± 3 days, Day 42 ± 3 days
  Patients were asked if they were going back to work.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, Prof. Dr. med., Principal Investigator — Emergency Department University Hospital Basel
Locations (1):
- Emergency Department University Hospital Basel, Basel, Switzerland